CLINICAL TRIAL: NCT05369975
Title: A Controlled, Open-label PA Efficacy and Safety Study in Imlifidase Desensitised Kidney Tx Patients With Positive XM Against a Deceased Donor Prior to Imlifidase Treatment, Including Non-comparative Registry and Concurrent Reference Cohorts
Brief Title: Efficacy and Safety in Imlifidase Desensitized Kidney Tx Patients, Including Two Non-Comparative Reference Cohorts
Acronym: PAES
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-HMedIdeS-19; 2021-002640-70 (EudraCT Number)
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplantation in Highly Sensitized Patients
Keywords: Desensitization; Highly sensitized; Positive crossmatch; Unlikely to be transplanted; Renal transplantation; Kidney transplantation; Deceased donor; End-Stage Renal Disease; ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Mac-1-like protein, Streptococcus

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomised trial in highly sensitized adult kidney transplant patients with positive XM against an available deceased donor.
  The rational for a non-randomised trial is that no other effective or approved desensitization protocol exists in deceased-donor kidney transplantation that would provide a suitable control.
  A non-comparative concurrent reference cohort from participating sites will be included to address differences in-site practice and experience.
  A non-comparative historical reference cohort from the CTS registry will be included to address the outcome in a less sensitized patient group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Imlifidase (Experimental): Imlifidase, is provided as a freeze-dried powder for concentrate for solution for infusion, 11 mg per vial. After reconstitution with sterile water for injection, the concentrate contains 10 mg/mL imlifidase. Imlifidase is administered intravenously as one infusion of 0.25 mg/kg over 15 minutes within 24 hours prior to transplantation. A second dose of 0.25 mg/kg may be given if the first imlifidase dose is considered not to have had sufficient effect. The second dose can be administered within 24 hours after the first dose.
  Interventions: Drug: Imlifidase
- Non-Comparative Concurrent Reference Cohort (Other): Patients in the non-comparative prospective concurrent reference cohort (with any grade of sensitization and negative XM) will receive medications, both pre- and post-transplant, in accordance with each clinic's routine for kidney transplanted patients.
  Interventions: Other: Normal Transplantation Routine
- Non-Comparative Historical Reference Cohort (Other): Patients in the non-comparative historical reference cohort (with less sensitization and negative XM) randomly selected from the CTS registry have been transplanted and treated in accordance with standard-of-care for kidney transplanted patients. Patients transplanted in 2010 and onwards will be selected to optimize the probability that these patients will have received about the same maintenance immunosuppressive treatment as the patients in the current trial will receive.
  Interventions: Other: Normal Transplantation Routine

INTERVENTIONS:
Drug: Imlifidase — Imlifidase is an immunoglobulin G (IgG)-degrading enzyme of Streptococcus pyogenes that is highly selective towards IgG. The cleavage of IgG generates one F(ab')2- and one homodimeric Fc-fragment and efficiently neutralizes Fc-mediated activities of IgG.
  Other Names: IdeS, HMED-IdeS
  Arms: Imlifidase
Other: Normal Transplantation Routine — Transplantation and pre- and post-transplantation therapies in accordance with the clinic's normal transplantation routine.
  Arms: Non-Comparative Concurrent Reference Cohort; Non-Comparative Historical Reference Cohort

SUMMARY:
An open-label post authorization efficacy and safety study evaluating graft failure-free survival at 1-year in highly sensitized end-stage renal disease (ESRD) patients with positive crossmatch (XM) against a deceased donor prior to desensitized with imlifidase and subsequent kidney transplantation. Two non-comparative reference cohorts are included to assess the impact of differences in post-transplantation management and outcome in less sensitized patients.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo pre-screening to determine eligibility for study entry. All highly sensitized ESRD patients with a positive XM will be desensitized with imlifidase to convert the XM to negative and then transplanted. Following transplantation, patients will receive induction therapies (corticosteroids, rabbit anti-human thymocyte immunoglobulin (rATG)), rejection prophylaxis (high-dose intravenous immunoglobulin (IVIg), rituximab or biosimilar) and maintenance immunosuppressive therapies. The patients will be followed for 12 months.

The efficacy of imlifidase per se, i.e. rapidly cleavage of IgG to enable transplantation, is not reflected by the important clinical outcomes 1-year graft failure-free survival and kidney function. These are instead a measure of effectiveness and safety in the real-world transplantation setting. It should be noted that patient outcome is highly dependent on the post-transplantation management, as well as compliance to maintenance immunosuppressive therapy.

All patients with donor specific antibodies (DSAs) are at risk for antibody-mediated reactions (AMRs). Imlifidase removes DSA quickly and efficiently at the time of transplantation but, as with other desensitization methods, the antibodies are expected to re-occur after transplantation. The highly sensitized patients included in this trial must therefore be closely monitored for any signs of AMR. Protocol kidney biopsies will be performed at 6 months and 1 year after transplantation. For-cause biopsies, DSA and estimated glomerular filtration rate (eGFR) will be collected to assess AMR frequency.

A non-comparative concurrent reference cohort consisting of kidney transplanted patients from participating trial sites with any grade of sensitization and a negative XM towards their donor will be included in the trial to address differences in-site practice, experience, and amount of immunosuppressive therapies given that may have an impact on the overall results for the imlifidase-treated cohort. Once a highly sensitized imlifidase treated patient has been transplanted at a site, subsequent patients who are offered a compatible kidney will be offered the opportunity to be included in the trial as part of the reference cohort group and transplanted. The goal is to have at least 1 or 2 patients from each site participating in the non-comparative concurrent reference cohort. Given that the patients in this cohort will be qualitatively different from the imlifidase treated patients, formal statistical comparisons will not be appropriate. Patients included in the non-comparative concurrent reference cohort will be followed for 12 months after transplantation and treated in accordance with each clinic's normal transplantation routines.

A second, non-comparative historical reference cohort of 100 kidney transplanted patients will be randomly selected from the Collaborative Transplant Study (CTS) registry in accordance with the inclusion and exclusion criteria provided in the protocol prior to commencement of the active trial. No clinical activities will be done to this historical reference cohort. The patients of this cohort will be less sensitized compared to the imlifidase-treated cohort, have a negative XM towards their donor and have been transplanted during 2010 or later. Since patients in this cohort are expected to have both a better prognosis and a higher graft survival rate at 1 year than the imlifidase-treated patients, formal statistical comparison between the groups would be inappropriate. The year 2010 was chosen as cut-off for inclusion in the non-comparative historical reference cohort to make it likely that the patients in this group have received the same maintenance immunosuppression as is given today to most kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for ALL patients

1. Male or female patient aged 18-75 years
2. ABO-compatible deceased donor aged 10-70 years

Inclusion criteria for IMLIFIDASE patients

1. ESRD active on the renal transplant waiting list of a kidney allocation system at the time of screening
2. High sensitization with the highest unmet medical need unlikely to be transplanted under the available kidney allocation system including prioritisation programmes for highly sensitized patients
3. Known DSA against an available deceased donor
4. Positive crossmatch test determined by complement-dependent cytotoxicity crossmatch (CDCXM) and/or flow cytometric crossmatch (FCXM) against an available deceased donor. If physical XM tests are not practically possible due to lack of time, patients may be included on a virtual crossmatch (vXM) predictive of a positive XM test.
5. Signed Informed Consent obtained before any trial-related procedures
6. Willingness and ability to comply with the protocol

Inclusion criteria for patients in the NON-COMPARATIVE CONCURRENT REFERENCE COHORT

1. Active on the renal transplant waiting list at a participating trial site at the time of screening
2. An acceptable kidney transplant from a deceased donor
3. Signed Informed Consent obtained before any trial related procedures
4. Willingness and ability to comply with the protocol

Inclusion criteria for patients in the NON-COMPARATIVE HISTORICAL REFERENCE COHORT

1. ESRD with a kidney transplant from a deceased donor
2. Being transplanted in Europe after 01-Jan-2010 and included in the CTS registry
3. Panel reactive antibodies (PRA) ≥ 50% (CDC T- or B-cell PRA, calculated panel reactive antibodies (cPRA), or virtual panel reactive antibodies (vPRA))
4. Maintenance immunosuppression (intention to treat) with calcineurin inhibitor, mycophenolate mofetil (MMF) and corticosteroids in combination

Exclusion Criteria:

Exclusion criteria for IMLIFIDASE patients and for patients in the NON-COMPARATIVE CONCURRENT REFERENCE COHORT

1. Use of investigational agents within 5 terminal elimination half-lives prior to the transplantation
2. Malignancy within 5 years prior to transplantation
3. Positive serology for human immunodeficiency virus (HIV)
4. Clinically relevant active infection(s) as judged by the investigator
5. Contemporaneous participation in medical device studies
6. Known mental incapacity or language barriers precluding adequate understanding of the Informed Consent information and the trial activities
7. Inability by the judgement of the investigator to participate in the trial for any other reason

Exclusion criteria for IMLIFIDASE patients

1. Previous treatment with imlifidase
2. Previous high dose IVIg treatment (2 g/kg) within 28 days prior to imlifidase treatment
3. Positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test
4. Breast feeding or pregnancy
5. Hypersensitivity to the active substance (imlifidase) or to any of the excipients
6. Ongoing serious infections
7. Present, or history of, thrombotic thrombocytopenic purpura (TTP), or known familial history of TTP
8. Severe other condition requiring treatment and close monitoring e.g. cardiac failure ≥ grade 4 (New York Heart Association), unstable coronary disease or oxygen dependent respiratory disease
9. Female of childbearing potential, not willing to use effective contraception during the 3 weeks following treatment with imlifidase. In the context of this trial, an effective method is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly such as:

   1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation; (i) oral, (ii) intravaginal, or (iii) transdermal
   2. progestogen-only hormonal contraception associated with inhibition of ovulation; (i) oral, (ii) injectable, or (iii) implantable
   3. intrauterine device (IUD)
   4. intrauterine hormone-releasing system (IUS)
   5. bilateral tubal occlusion
   6. vasectomised partner
   7. true abstinence: When this is in line with the preferred and usual lifestyle of the patient. [Periodic abstinence (such as calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception]
10. Any other reason that, in the view of the investigator, precludes transplantation

Exclusion criteria for patients in the NON-COMPARATIVE HISTORICAL REFERENCE COHORT

1. Patients treated with mammalian target of rapamycin (mTOR) inhibitors
2. Patients treated with belatacept

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Graft failure-free survival 1 year after transplantation following imlifidase treatment | 12 months after transplantation
  Graft failure is defined as permanent return to dialysis for at least 6 weeks, re-transplantation, or nephrectomy. Patients who die from any cause will be considered as having graft failure.
  If a patient is not undergoing transplantation following imlifidase treatment the patient will be censored at time zero when constructing Kaplan-Meier curves for graft failure-free survival.
  The 1-year graft failure-free survival rates will be extracted from Kaplan-Meier curves.
  Time from enrolment to the first of death or graft failure will be used as time variable.

SECONDARY OUTCOMES:
Graft failure-free survival 1 year after transplantation in non-comparative concurrent reference cohort | 12 months after transplantation
  Graft failure is defined as permanent return to dialysis for at least 6 weeks, re-transplantation, or nephrectomy. Patients who die from any cause will be considered as having graft failure.
  The 1-year graft failure-free survival rates will be extracted from Kaplan-Meier curves.
  Time from enrolment to the first of death or graft failure will be used as time variable.
Renal function up to 1 year after transplantation | Screening, pre-imlifidase, 24, 48 and 72 hours, Days 5, 6, 8, 10 and 15, at 1, 3 and 6 months and at 1 year
  Renal function will be assessed at several timepoints for the imlifidase-treated cohort, the non-comparative concurrent reference cohort and the non-comparative historical reference cohort. Of note, less frequent sampling is done to the non-comparative concurrent reference cohort as compared with the imlifidase treatment group. For the historical reference cohort kidney function will be measured by serum/plasma creatinine category at 3 and 6 months and 1 year (130 µmol/L, 130-259 µmol/L, 260-400 µmol/L and >400 µmol/L). eGFR will be available only in selected patients in the historical control cohort.
  eGFR is a measure of kidney function. The serum/plasma creatinine levels will be analysed and eGFR will be calculated according to the modification of diet in renal disease (MDRD) equation.
  Reduced kidney function is characterised by a decreased eGFR value. eGFR will be set to 0 for patients treated with imlifidase who are not successfully transplanted.
Patient survival at 1 year after transplantation | 12 months after transplantation
  Patient survival will be assessed for the imlifidase-treated cohort, the non-comparative concurrent reference cohort and the non-comparative historical reference cohort.
  The 1-year patient survival rates will be extracted from Kaplan-Meier curves.
Graft survival at 1 year after transplantation | 12 months after transplantation
  Graft survival will be assessed for the imlifidase-treated cohort, the non-comparative concurrent reference cohort and the non-comparative historical reference cohort.
  Graft survival will be presented with Kaplan-Meier curves. Graft failure is defined as permanent return to dialysis for at least 6 weeks, re-transplantation, or nephrectomy. Patients who die will be censored at time of death.
Proportion of patients with conversion of a positive XM test to negative within 24 hours after imlifidase treatment | Pre-imlifidase, 2, 4 and 24 hours post-imlifidase.
  This outcome is applicable for the imlifidase-treated cohort only. XM testing will be performed using CDCXM and FCXM (B- and T-cells). If any of the B- or T-cells or both are positive, the patient is categorised as having a positive XM test.
HLA/DSA antibody levels up to 1 year after imlifidase treatment | Screening, pre-imlifidase, at 2, 4, 24, 48 and 72 hours, at Days 5, 6, 8, 15, at 1, 3 and 6 months, and at 1 year
  This outcome will be assessed for the imlifidase-treated cohort only. HLA antibodies will be analysed throughout the study using an IgG single antigen solid-phase immunoassay for class I and class II (SAB-HLA).
  Donor specific antibodies (DSAs) are identified by using the human leukocyte antigen (HLA) profile data from the donor and the recipient to identify HLA-mismatches.
  Antibodies directed against donor HLA with levels >1000 mean fluorescence intensity (MFI) prior to imlifidase infusion are considered pre-transplant DSAs. The MFIs will be summarized for all DSAs with an MFI of ≥1000 at any time during the trial.
Imlifidase pharmacokinetics (AUC) | Pre-imlifidase, 30 minutes and 2, 4, 8, 24, 48 and 72 hours, Days 5, 6, 8, 10, and 15
  AUC = Area under the imlifidase plasma concentration versus time curve Sampling for pharmacokinetic (PK) analyses will be performed for a subgroup of about 20 imlifidase treated patients at a selected number of sites.
Imlifidase pharmacokinetics (Cmax) | Pre-imlifidase, 30 minutes and 2, 4, 8, 24, 48 and 72 hours, Days 5, 6, 8, 10, and 15
  Cmax = Maximum observed plasma concentration of imlifidase following dosing. Sampling for PK analyses will be performed for a subgroup of about 20 imlifidase treated patients at a selected number of sites.
Imlifidase pharmacokinetics (tmax) | Pre-imlifidase, 30 minutes and 2, 4, 8, 24, 48 and 72 hours, Days 5, 6, 8, 10, and 15
  tmax = Time point for maximum observed plasma concentration of imlifidase following dosing.
  Sampling for PK analyses will be performed for a subgroup of about 20 imlifidase treated patients at a selected number of sites.
Imlifidase pharmacokinetics (t1/2) | Pre-imlifidase, 30 minutes and 2, 4, 8, 24, 48 and 72 hours, Days 5, 6, 8, 10, and 15
  t1/2 = Terminal half-life of imlifidase Sampling for PK analyses will be performed for a subgroup of about 20 imlifidase treated patients at a selected number of sites.
Imlifidase pharmacokinetics (CL) | Pre-imlifidase, 30 minutes and 2, 4, 8, 24, 48 and 72 hours, Days 5, 6, 8, 10, and 15
  CL = Clearance of imlifidase. Sampling for PK analyses will be performed for a subgroup of about 20 imlifidase treated patients at a selected number of sites.
Imlifidase pharmacokinetics (Vz) | Pre-imlifidase, 30 minutes and 2, 4, 8, 24, 48 and 72 hours, Days 5, 6, 8, 10, and 15
  CL = Clearance of imlifidase. Sampling for PK analyses will be performed for a subgroup of about 20 imlifidase treated patients at a selected number of sites.
Imlifidase pharmacodynamics | Pre-imlifidase, 30 minutes and 2, 4, 8, 24, 48 and 72 hours, Days 5, 6, 8, and 10
  IgG concentration in patient serum will be measured. Composition of IgG fragments will be analysed and scored.
  Sampling for pharmacodynamic (PD) analyses will be performed for a subgroup of about 20 imlifidase treated patients at a selected number of sites.
Anti-drug antibodies (ADA) levels up to 1 year after imlifidase treatment | Days 8, and 15, at 1, 3 and 6 months, and at 1 year
  This outcome is applicable for the imlifidase-treated cohort only. Determination of anti-imlifidase IgG (ADA) concentration in serum will be performed centrally using a customised ImmunoCAP.
Frequency of delayed graft function (DGF) | Up to 7 days after transplantation
  Delayed graft function (DGF) will be assessed for the imlifidase-treated cohort and the non-comparative concurrent reference cohort.
  DGF is defined as need for dialysis within 7 days of transplantation.
Proportion of patients with biopsy- and serology (DSA)-confirmed antibody-mediated rejections (AMRs) | Up to 12 months after transplantation
  Frequency of AMRs will be assessed for the imlifidase-treated cohort and the non-comparative concurrent reference cohort.
  This includes protocol biopsies at 6 months and 1 year after transplantation in the imlifidase treatment group. For-cause biopsies will be obtained to confirm diagnosis for suspected AMRs in both treatment arms.
  All kidney biopsies (protocol and for-cause) in both cohorts will be evaluated according to Banff criteria version 2017 or later.
  DSA and eGFR will be analysed centrally for the imlifidase group and locally for the concurrent reference cohort.
Proportion of patients with biopsy- and serology (DSA)-confirmed cell-mediated rejections (CMRs) | Up to 12 months after transplantation
  Frequency of CMRs will be assessed for the imlifidase-treated cohort and the non-comparative concurrent reference cohort.
  This includes protocol biopsies at 6 months and 1 year after transplantation in the imlifidase treatment group. For-cause biopsies will be obtained to confirm diagnosis for suspected AMRs in both treatment arms.
  All kidney biopsies (protocol and for-cause) in both cohorts will be evaluated according to Banff criteria version 2017 or later.
  DSA and eGFR will be analysed centrally for the imlifidase group and locally for the concurrent reference cohort.
Proportion of patients with infusion-related reactions within 48 hours of imlifidase infusion | Up to 48 hours after transplantation
  This outcome is applicable for the imlifidase-treated cohort only. Infusion-related reactions that occurs within 48 hours of imlifidase treatment are considered adverse events of special interest (AESI).
Proportion of patients with severe or serious infections within 30 days after transplantation | Up to 30 days after transplantation
  This outcome will be assessed for the imlifidase-treated cohort and the non-comparative concurrent reference cohort.
  Severe or serious infections within 30 days after transplantation are considered AESI for both these cohorts.
Change in patient-reported life participation | Screening and at 1 year
  This outcome will be assessed for the imlifidase-treated cohort and the non-comparative concurrent reference cohort.
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Social Health domain "Ability to participate in social roles & activities" Short Form 8a will be used as a measure of the patients' health related quality of life.
  The questionnaire includes 8 questions about a persons ability to participate in different social activities and there are 5 different answers to choose from for each question: Never/Rarely/Sometimes/Usually/Always
Proportion of patients with rejection episodes (AMRs and CMRs) during the first post-transplant year in patients with a functioning graft at the end of the first post-transplant year | From transplantation to 1 year
  This outcome will be assessed for the non-comparative historical reference cohort only.
  Data for AMR/CMR rejection episodes during the first post-transplant year will be collected from the CTS registry.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Hansa Biopharma AB
Locations (22):
- Medizinische Universitaet Wien, Vienna, Austria
- UZ Leuven - Campus Gasthuisberg, Leuven, Belgium
- Institut klinicke a experimentalni mediciny (IKEM), Prague, Czechia
- France (3):
  - Centre Hospitalier Universitaire (CHU) de Rouen - Hôpital de Bois-Guillaume, Bois-Guillaume
  - CHU de Grenoble - Hôpital Michallon, La Tronche
  - Hôpital Necker - Enfants Malades, Paris
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum rechts der Isar der Technische Universitaet Muenchen, Munich
- Italy (2):
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero - Universitaria di Parma, Parma
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Erasmus University Medical Center, Rotterdam
- Department of Nephrology , Zaloška 7, Ljubljana, Slovenia
- Spain (4):
  - Hospital Del Mar, Servicio de Nefrología, Barcelona
  - Hospital Clínic de Barcelona, Unidad de Trasplante Renal, Barcelona
  - Vall d'Hebron University Hospital (HUVH), Barcelona
  - Hospital 12 de Octubre, Madrid
- Sweden (2):
  - Karolinska University Hospital, Huddinge
  - Uppsala University Hospital, Uppsala
- United Kingdom (2):
  - St. James University Hospital, Leeds
  - Leicester General Hospital, Leicester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vo A, Ammerman N, Jordan SC. New Therapies for Highly Sensitized Patients on the Waiting List. Kidney360. 2024 Aug 1;5(8):1207-1225. doi: 10.34067/KID.0000000000000509. Epub 2024 Jul 12. PMID 38995690